CLINICAL TRIAL: NCT02561299
Title: Orbital Vessel PreparaTIon to MaximIZe Dcb Efficacy in Calcified Below the Knee (BTK) Lesions - A Pilot Study
Acronym: OPTIMIZE BTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0007-P
Record Dates: First submitted 2015-08-26; First posted 2015-09-28 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: PAD; Vascular Calcification
Keywords: Drug-coated Balloons; Calcified Lesions; Orbital Atherectomy; Below the Knee; Paclitaxel; Lutonix 014 Drug-coated Balloon
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- OA with adjunctive DCB angioplasty (Experimental): Lesion preparation with Peripheral Orbital Atherectomy System followed by drug-coated balloon angioplasty
  Interventions: Device: Peripheral Orbital Atherectomy System; Device: 014 Drug Coated Balloon
- DCB angioplasty (Active Comparator): 014 Drug Coated Balloon angioplasty
  Interventions: Device: 014 Drug Coated Balloon

INTERVENTIONS:
Device: Peripheral Orbital Atherectomy System — Orbital Atherectomy
  Arms: OA with adjunctive DCB angioplasty
Device: 014 Drug Coated Balloon — Drug Coated Balloon

SUMMARY:
The purpose of this study is to prospectively evaluate acute and long term clinical results of orbital atherectomy (OA) with adjunctive drug coated balloon (DCB) angioplasty versus DCB angioplasty alone for treatment of Peripheral Artery Disease (PAD) in below the knee (BTK) lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age ≥ 18 years
* Rutherford Clinical Category 3 - 5
* Lesions [except in-stent restenosis (ISR)] of the distal popliteal (POP segment below the anatomical knee joint), anterior tibial, posterior tibial, tibial peroneal trunk, and peroneal arteries with ≥ 70 % diameter stenosis (DS) by angiography
* Presence of clearly visible calcification in two views (both sides of vessel at the same location) evaluated angiographically- [Computerized tomography (CT) angio images may substitute to confirm distribution of calcium, if available as standard of care]
* Length of calcium ≥ 25 % of total lesion length or ≥ 2 cm total length
* Target lesion length up to 20 cm

Exclusion Criteria:

* Subject or subject's legal representative is not willing to sign an Ethics Committee approved informed consent form or comply with the study protocol requirements
* Contraindicated by either device, per Instructions For Use
* Presence of inflow lesion (≥ 50 % DS) or inflow not successfully treated (≥ 50% DS and/or unresolved significant angiographic complication)
* Compromised outflow distal to the target lesion (≥ 70 % DS) or presence of lesion(s) or occlusion(s) located from 5 cm above the ankle to below the ankle joint space
* Subject has more than 2 target vessels requiring treatment
* The guide wire cannot be passed across the target lesion(s) and/or guide wire position distal to target lesion(s) outside vessel lumen
* Presence of significant (≥ 70 % DS) lesion(s) or occlusion(s) not meeting the study criteria which were not successfully treated during the index procedure (≥ 50 % DS and/or significant angiographic complication)
* Subject has planned amputation (including minor) of the index limb or previous major amputation of the contralateral limb
* Creatinine > 2.5 mg/dL, unless on dialysis
* Subject has any significant medical condition which, in the Investigator's opinion, may interfere with the subject's optimal participation in the study
* Subject is participating in an investigational drug or device study that has the potential to clinically interfere with the study outcome measures
* Subject is pregnant or planning to become pregnant within the study period
* Subject has an unresolved severe systemic infection
* Subject has an anticipated life span of less than one year
* Subjects with known hypersensitivity to paclitaxel or paclitaxel related compounds
* Subjects who cannot receive recommended anti-platelet and/or anticoagulant therapy
* Pre-dilatation of the target lesion prior to randomization and OA treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Marianne Brodmann, Dr., Principal Investigator — Medical University of Graz, Austria; Professor Gunnar Tepe, Dr., Principal Investigator — Klinikum Rosenheim Germany; Professor Thomas Zeller, Dr., Principal Investigator — Herz-Zentrum Bad Krozingen Germany
Locations (7):
- Austria (2):
  - Medical University of Graz, Graz
  - Vascular Clinic - Hanusch Hospital, Vienna
- Germany (5):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Fürst-Strium-Klinik Bruchsal, Bruchsal
  - SRH Klinikum Karlsbad- Langensteinbach GmbH, Langensteinbach
  - Universität Leipzig, Leipzig
  - Romed Klinikum Rosenheim, Rosenheim

REFERENCES:
- [Result] Zeller T, Giannopoulos S, Brodmann M, Werner M, Andrassy M, Schmidt A, Blessing E, Tepe G, Armstrong EJ. Orbital Atherectomy Prior to Drug-Coated Balloon Angioplasty in Calcified Infrapopliteal Lesions: A Randomized, Multicenter Pilot Study. J Endovasc Ther. 2022 Dec;29(6):874-884. doi: 10.1177/15266028211070968. Epub 2022 Jan 27. PMID 35086385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Started | 32 | 34
Completed | 27 | 28
Not Completed | 5 | 6
Not completed — Death | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8.5) | 76.5 (7.1) | 75.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 26 | 25 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Rutherford Clinical Category [Count of Participants; unit: Participants]
  Severe Claudication (3) | 10 | 8 | 18
  Ischemic Rest Pain (4) | 2 | 4 | 6
  Minor Tissue Loss (5) | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Device Success
Description: Device success was defined as the ability to achieve successful delivery and deployment of the drug-coated balloon (DCB) to the target lesion as described per Instructions for Use (IFU) within 3 minutes of insertion without removal and use of an additional device. The percentage of success was based on the number of DCB devices used.
Time Frame: During the procedure
Measure: Count of Units; unit: Drug Coated Balloons
Units Other Than Participants: Drug Coated Balloons
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Number analyzed (Participants) | 32 | 34
Number analyzed (Drug Coated Balloons) | 45 | 48
Drug Coated Balloons | 42 | 39

2. Primary Outcome: Patency of the Target Lesion at 6 Months and 12 Months Post-Procedure
Description: Patency of the target lesion as reported by the Duplex Ultrasound (DUS) Core Laboratory. Vessel patency at 6 months and 12 months by Duplex Ultrasound (DUS), where patency is defined as <50% restenosis within the treated lesion area. Patency was assessed by the DUS Core Laboratory.
Time Frame: 6 months and 12 months post-procedure
Population: Lesions with available data for patency assessment by the DUS Core Lab
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Number analyzed (Participants) | 32 | 34
Number analyzed (Lesions) | 35 | 37
Lesions
  Patency at 6 months: number analyzed (Participants) | 16 | 9
  Patency at 6 months: number analyzed (Lesions) | 17 | 10
  Patency at 6 months | 15 | 5
  Patency at 12 months: number analyzed (Participants) | 16 | 10
  Patency at 12 months: number analyzed (Lesions) | 17 | 11
  Patency at 12 months | 15 | 6

3. Primary Outcome: Freedom From Clinically-Driven Target Lesion Revascularization (CD-TLR) at 6 Months and 12 Months Post-Procedure
Description: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant was free from CD-TLR through 6 months and 12 months.
Time Frame: 6 months and 12 months post-procedure
Measure: Number (95% Confidence Interval); unit: % probability
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Number analyzed (Participants) | 32 | 34
% probability
  Freedom from CD-TLR at 6 months | 96.8 [90.6 to 103.0] | 94.1 [86.2 to 102.0]
  Freedom from CD-TLR at 12 months | 86.4 [74.0 to 98.8] | 91.0 [81.2 to 100.7]

4. Primary Outcome: Freedom From Unplanned, Unavoidable Major Amputation of the Index Limb at 6 Months and 12 Months Post-Procedure
Description: A Kaplan-Meier analysis was performed to determine the percent probability that the study participant was free from an unplanned, unavoidable major amputation of the index limb through 6 months and 12 months.
Time Frame: 6 months and 12 months post-procedure
Measure: Number (95% Confidence Interval); unit: % probability
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Number analyzed (Participants) | 32 | 34
% probability
  Freedom from major amputation at 6 months | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]
  Freedom from major amputation at 12 months | 96.6 [89.9 to 103.2] | 100.0 [100.0 to 100.0]

5. Primary Outcome: Freedom From Major Adverse Events (MAEs) at 6 Months and 12 Months Post-Procedure
Description: A Kaplan-Meier analysis was performed to determine the percent probability that the study participant was free from a major adverse event (MAE) through 6 months and 12 months. Major adverse events were defined as: clinically-driven target lesion revascularization (CD-TLR); unplanned, unavoidable major amputation of the index limb; and death within 30 days of the index procedure.
Time Frame: 6 months and 12 months post-procedure
Measure: Number (95% Confidence Interval); unit: % probability
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Number analyzed (Participants) | 32 | 34
% probability
  Freedom from MAE at 6 months | 90.6 [80.5 to 100.7] | 91.2 [81.6 to 100.7]
  Freedom from MAE at 12 months | 77.7 [63.1 to 92.3] | 85.3 [73.4 to 97.2]

6. Primary Outcome: Change in Rutherford Category at 6 Months and 12 Months Post-Procedure
Description: Rutherford Classification (RC) is a commonly used clinical grading system for describing peripheral arterial disease (PAD) on a scale of 0 to 6. RC 6 is the most severe form of PAD.
  There are seven Rutherford categories used to grade the severity of peripheral artery disease; 0: asymptomatic, 1: mild claudication, 2: moderate claudication, 3: severe claudication, 4: ischemic rest pain, 5: minor tissue loss, 6: major tissue loss.
  The change in Rutherford category is presented as the distribution at baseline compared to that at 6- and 12-months post-procedure.
Time Frame: Baseline, 6 months and 12 months post-procedure
Population: The number of participants analyzed at 6 and 12 months differs from the overall number due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
Number analyzed (Participants) | 32 | 34
Participants
  Baseline: Rutherford Category 0 | 0 | 0
  Baseline: Rutherford Category 1 | 0 | 0
  Baseline: Rutherford Category 2 | 0 | 0
  Baseline: Rutherford Category 3 | 10 | 8
  Baseline: Rutherford Category 4 | 2 | 4
  Baseline: Rutherford Category 5 | 20 | 22
  Baseline: Rutherford Category 6 | 0 | 0
  6 months: number analyzed (Participants) | 22 | 17
  6 months: Rutherford Category 0 | 6 | 7
  6 months: Rutherford Category 1 | 5 | 1
  6 months: Rutherford Category 2 | 2 | 0
  6 months: Rutherford Category 3 | 1 | 1
  6 months: Rutherford Category 4 | 0 | 0
  6 months: Rutherford Category 5 | 8 | 8
  6 months: Rutherford Category 6 | 0 | 0
  12 months: number analyzed (Participants) | 24 | 18
  12 months: Rutherford Category 0 | 10 | 8
  12 months: Rutherford Category 1 | 3 | 3
  12 months: Rutherford Category 2 | 2 | 1
  12 months: Rutherford Category 3 | 4 | 1
  12 months: Rutherford Category 4 | 0 | 0
  12 months: Rutherford Category 5 | 5 | 5
  12 months: Rutherford Category 6 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization through subject trial completion, up to 24 months.
Description: All serious adverse events were collected throughout the subject participation in the trial. Procedural complications were considered adverse events and were collected from randomization through discharge. Per the protocol, the Core Lab's final classification of endpoint events including Severe Dissection, Perforation, Distal Embolization, and Slow Flow/No Reflow is used for reporting purposes and may differ in classification from site reported adverse events.
Arm/Group | OA With Adjunctive DCB Angioplasty | DCB Angioplasty
All-Cause Mortality (participants affected / at risk) | 2/32 | 4/34
Serious Adverse Events (participants affected / at risk) | 29/32 | 22/34
Other Adverse Events (participants affected / at risk) | 4/32 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OA With Adjunctive DCB Angioplasty (N=32) | DCB Angioplasty (N=34)
Angina Pectoris (Ischemic Chest Pain) (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmias (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac/Cardiopulmonary Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Dysfunction-Acute Heart Failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Dysfunction-Chronic Heart Failure or Aggravated (Cardiac disorders) | 2 (3) | 5 (5)
Cardiac Valve Disorders (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac-Other (Cardiac disorders) | 1 (1) | 0 (0)
New/Worsening Infection (Vascular disorders) | 10 (16) | 5 (10)
New/Worsening Pain (Vascular disorders) | 6 (7) | 2 (2)
New/Worsening Wound (Vascular disorders) | 8 (17) | 8 (13)
Peripheral Artery Restenosis (Vascular disorders) | 4 (6) | 6 (9)
Peripheral Artery Stenosis (Vascular disorders) | 5 (6) | 8 (9)
Peripheral Thrombus/Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral Artery Psedoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral Artery Thrombus/Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bleeding/Hemorrhage,Access Site (Vascular disorders) | 1 (1) | 0 (0)
Bleeding/Hemorrhage, Non Access Site (Vascular disorders) | 2 (2) | 0 (0)
Carotid Artery Disease (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 1 (2)
Gastrointestinal Infection/Inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic/Biliary System Disorders (e.g liver, bile duct) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Digestive Disorders-Other (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chronic Mental Illness (e.g. anxiety, depression) (Psychiatric disorders) | 1 (1) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 4 (4) | 0 (0)
Syncope/Loss of Consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (2) | 1 (1)
Chronic Renal Failure or Worsened (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 3 (3) | 1 (2)
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory/Thoracic Disorders-Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Blood and Lymphatic System Disorder-Anemia (General disorders) | 1 (1) | 1 (1)
Blood and Lymphatic System Disorders-Other (General disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 1 (1) | 2 (3)
Chest Pain, Non-Cardiac (General disorders) | 0 (0) | 1 (1)
Chest Pain, Unspecified (General disorders) | 1 (1) | 0 (0)
Endocrine/Metabolic Disorders (General disorders) | 1 (2) | 2 (2)
Infection-Other-Localized (General disorders) | 1 (1) | 1 (1)
Infection-Systemic (General disorders) | 2 (3) | 1 (1)
Injury/Trauma (General disorders) | 3 (3) | 4 (4)
Multi-Organ Failure (General disorders) | 0 (0) | 2 (2)
Pain-Other (General disorders) | 0 (0) | 1 (1)
Perhipheral Edema (General disorders) | 0 (0) | 1 (1)
Shock (General disorders) | 1 (1) | 0 (0)
Sleep Disorders (General disorders) | 0 (0) | 1 (1)
Adverse Event-Other (General disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OA With Adjunctive DCB Angioplasty (N=32) | DCB Angioplasty (N=34)
Peripheral Artery Perforation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Peripheral Artery Thrombus/Thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood and Lymphatic System Disorder-Anemia (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT02561299/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT02561299/SAP_001.pdf